CLINICAL TRIAL: NCT01982279
Title: One Year Change in Caloric Compensation and Eating in the Absence of Hunger in French Preschool Children
Brief Title: Longitudinal Measurement of Caloric Compensation and Eating in the Absence of Hunger in French Preschool Children
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: European Union (Other)
Responsible Party: Sponsor
Other Study IDs: HabEat WP31 Follow up; INRA WP31 FU; WP31.FU. INRA (Other: INRA)
Record Dates: First submitted 2013-10-30; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Caloric compensation; Eating in the absence of hunger; Preschool children; Maternal feeding practices; Maternal eating behavior; one year; children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objectives: The aims were to measure one year change in caloric compensation (CC) and eating in the absence of hunger (EAH) in 3 to 6 year-old French children in their regular eating context and to link these change with individual characteristics (adiposity, age, gender) and maternal feeding practices.

Three series of measurements of caloric compensation (CC) and eating in the absence of hunger (EAH) were conducted: at baseline, and 3 (FU3M) and 15 (FU15M) months later. Each serie of measurement was composed of three consecutive weeks an identical lunch was served in four preschool canteens reaching 236 children. The first lunch was a control session. For the CC situation (week 2), thirty minutes before the lunch children were offered a preload (137 kcal). For the EAH situation (week 3), ten minutes after lunch children were exposed to palatable foods (430 kcal). Food intake was measured at the individual level. Maternal eating behaviour and feeding practices were measured by questionnaires. Child's height and weight were measured by a medical doctor.

ELIGIBILITY:
Inclusion Criteria:

* To be registered to the school canteen, to provide parental approval at inclusion and at the FU15M

Exclusion Criteria:

* Chronic disease or food allergies

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population was composed of 236 children at inclusion. Among them, 98 participated in the three time of measurements of caloric compensation or eating in the absence of hunger.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2011-02; Primary Completion 2011-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in caloric compensation in 15 months | one week
  To evaluate the change in caloric compensation across time, caloric compensation was measured at baseline, 3 and 15 months after baseline, in the same conditions. At each time point to assess caloric compensation, children were offered a chocolate bun 30 minutes before the lunch. The food intake at lunch was recorded. We calculated if children compensated the chocolate bun, by comparing energy intake at this lunch with energy intake from a control lunch which took place one week before.
Control measurement of energy intake at baseline | One week
  We conducted a control lunch and recorded food intake of each child. This measurement was conducted a week before measuring caloric compensation.
Change in eating in the absence of hunger in 15 months | one week.
  In order to evaluate the change in eating in the absence of hunger across time, a measurement was conducted at baseline, 3 months and 15 months after baseline. To collect the measurement of eating in the absence of hunger, we offered palatable foods to children 10 minutes after their lunch. We recorded the energy intake from these post-meal foods. At each time point, this measurement was conducted one week after the measurement of caloric compensation.
Control measurement of energy intake three months after baseline | One week
  We conducted a control lunch and recorded food intake of each child. This measurement was conducted a week before measuring caloric compensation.
Control measurement of energy intake fifteen months after baseline | One week
  We conducted a control lunch and recorded food intake of each child. This measurement was conducted a week before measuring caloric compensation.

SECONDARY OUTCOMES:
Maternal feeding practices and eating behavior | one month after inclusion
  Using a validated questionnaire, we collected information about maternal feeding practices (Comprehensive Feeding Practices Questionnaire, Musher-Eizenman & Holub, 2007) and eating behaviour (Dutch Eating Behaviour Questionnaire, Van Strien, 1986).

CONTACTS AND LOCATIONS:
Overall Officials: Nicklaus Sophie, phD, Principal Investigator — Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Locations (1):
- Centre des Sciences du Goût et de l'Alimentation, Dijon, France

REFERENCES:
- See also: Web site for the main research project funded by the European Union — http://www.habeat.eu/